CLINICAL TRIAL: NCT06331416
Title: Multiparametric Home Telemonitoring of Patients With Chronic Obstructive Pulmonary Disease Exacerbation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Confalonieri Marco, MD, MD, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEUR-2023-Em-145
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: COPD; COPD Exacerbation Acute
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Open-label randomized controlled trial, allocation ratio 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental)
  Interventions: Device: Telemonitoring
- Standard of care (No Intervention)

INTERVENTIONS:
Device: Telemonitoring — Patients will be asked to carry out one measurement (arterial pressure, oxygen saturation, body temperature, heart rate, spirometry) every 24 hours for 90 days. The system will be supplied by the company Vivisol. The telemonitoring data will be read once a day and the principal investigator will be alerted in case of alteration of any parameter. If vital parameters remain stable, a phone call will be performed every 5 days. In case of compromise of any parameter, the patient will be offered a phone call within the same day. In case of new occurrence of any respiratory or non-respiratory symptoms, the patient must contact the principal investigator and he will be offered a phone call or a video-assisted call within the same day. If the alterations or symptoms persist for 24 hours, or in any case upon decision of the investigator in charge, the patient will be offered an in-person evaluation in the same day. If deemed necessary according to usual care, the patient will be hospitalized.
  Arms: Telemonitoring

SUMMARY:
Chronic obstructive pulmonary disease (COPD) exacerbations are risk factors for disease progression and short-term re- hospitalizations. We propose a randomized controlled trial to evaluate the efficacy of a one-device multiparameter telemonitoring in reducing functional decline, symptoms, and risk of re-hospitalization of patients discharged after hospitalization for exacerbated COPD.

DETAILED DESCRIPTION:
Respiratory diseases such as asthma, chronic obstructive pulmonary disease (COPD), lung cancer, obstructive sleep apnea syndrome, pulmonary fibrosis and others are important causes of morbidity and mortality and have a substantial impact on healthcare costs. Furthermore, the Coronavirus-19 (COVID-19) pandemic has shown how respiratory complications are the most dangerous for infected subjects, as they can evolve into a severe pneumonia burdened by either subacute or chronic complications. Strict monitoring, early treatment initiation and timely hospitalization are fundamental to ameliorate short-term prognosis and reduce long-term sequelae of all acute respiratory conditions, including chronic obstructive pulmonary disease (COPD). Indeed, acute worsening of respiratory symptoms, called exacerbations, often occur during the course of the disease. COPD exacerbations are associated with an accelerated decline in respiratory function, and exacerbation frequency or intensity is a powerful predictor of future episodes and ultimate mortality which reaches as high as 50% at 5 years. Indeed, exacerbation frequency is the strongest single factor related to future exacerbations, and mortality rates increase 3-fold as exacerbation frequency increases from 0 to 3 or more per year. Recent data shown that 30-day readmission rate for COPD patients after discharge ranged from 22.6% to 24%, while 90-day readmission was 35.1% to 43% in different studies. Furthermore, severe COPD exacerbations resulting in hospitalization can be up to 60 times more expensive than mild or moderate exacerbations managed by primary care services. As a consequence, the medical community have launched numerous initiatives to reduce exacerbations, with a particular focus on reducing readmissions. These initiatives involve improving medication regimens and adherence, smoking cessation, pulmonary rehabilitation, assessments for oxygen supplementation and noninvasive ventilation, and close follow-up by clinicians following discharge. At the current state of things, patients discharged after an hospitalization for COPD exacerbation are followed-up through discrete, in-person, evaluation within one to three months. However, this timeframe is often not sufficient to identify clinical deterioration and the need for changes in the therapeutic strategy (e.g. switch of inhaler, counselling on the inhalation technique, need for oral add-on therapy) to avoid recurrence of symptoms and re-hospitalization. Nevertheless, there are no established programs to help medical doctors reduce COPD re-admissions. Since over two decades, telemedicine has been demonstrated effective in improving patients' health-related quality of life and in increasing the efficiency of care processes, but it has only recently been proposed as a strategy to reduce COPD readmission rate. Indeed, The COVID-19 pandemic has increased the awareness on the available systems for telemonitoring and favored the development of new ones. Telemonitoring is one major field of telemedicine which encompasses remote tracking of physiological parameters, either in real time or using store-and-forward technologies, allowing to screen for the patients who could benefit most of either home visits or hospitalization. Multiple devices have been made available for these purposes during the COVID-19 pandemic. We designed a randomized controlled trial to evaluate the ability of telemonitoring to avoid lung function decline, reduce symptoms and the risk of re-hospitalizations of patients discharged after a COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign the informed consent form.
2. Already established diagnosis of COPD according to Global Initiative for Obstructive Lung Disease (GOLD) guidelines.[13]
3. Diagnosis of COPD exacerbation at admission, according to GOLD guidelines.[13]
4. Arterial partial pressure of oxygen (PaO2) < 60 mmHg in ambient air at rest at admission and arterial partial pressure of oxygen (PaO2) > 60 mmHg in ambient air at rest at discharge, if not on long-term oxygen therapy on ventilation.
5. Arterial partial pressure of oxygen (PaO2) < 55 mmHg on usual oxygen supplement (L/min) and arterial partial pressure of oxygen (PaO2) > 60 mmHg on oxygen supplement at discharge, if already on long-term oxygen therapy on ventilation.

g) Age <= 90 and >= 18 years old at randomization.

Exclusion Criteria:

1. Heart failure as the main cause of acute respiratory failure
2. Acute pulmonary embolism/chronic pulmonary thromboembolism
3. Interstitial lung disease as the main cause of acute respiratory failure
4. Pneumonia as the main cause of acute respiratory failure
5. Chronic renal failure with dialysis dependence
6. Immunosuppression (i.e. cancer on treatment, post-organ transplantation, HIV-positive, on immunosuppressant therapy)
7. Progressive neuro-muscular disorders
8. Cognitively impaired, dementia or decompensated psychiatric disorder
9. Quadriplegia/Hemiplegia or quadriparesis/hemiparesis
10. Do-not-resuscitate order
11. Any other condition that in the opinion of the investigator may significantly impact with patient's capability to comply with the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization at 90 days | 90 days
  Proportion of re-hospitalized patients by day 90 in both groups

SECONDARY OUTCOMES:
Re-hospitalization at 30 days | 30 days
  Proportion of re-hospitalized patients by day 30 in both groups
Functional decline | 90 days
  Proportion of patients with ≥ 30 mL deflection in the predicted value of forced expiratory volume in the first second (FEV1) at spirometry or increase in COPD assessment test (CAT) score for symptoms evaluation ≥ 2 points between the first visit (one month after discharge) and the second visit (three months after discharge) in both groups.
Unplanned medical evaluations | 90 days
  Number of unplanned pneumological evaluation in both groups.
Need for mechanical ventilation at 30 days | 30 days
  Proportion of patients who require mechanical ventilation (either noninvasive or invasive) by day 30 in both groups.
Need for mechanical ventilation at 90 days | 90 days
  Proportion of patients who require mechanical ventilation (either noninvasive or invasive) by day 90 in both groups.
Satisfaction score | 90 days
  Self-reported score for overall satisfaction ≥ 8/10 for ≥ 80% of patients in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Confalonieri, MD, Study Chair — University of Trieste
Locations (1):
- SC Pneumologia, Azienda Sanitaria Universitaria Giuliano-Isontina, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon motivated request to the PI
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From the end of the study for 2 years
Access Criteria: email to the PI